CLINICAL TRIAL: NCT07065981
Title: Comparison of Upper Extremity Functional Exercise Capacity Between Lung Transplant Recipients and Healthy Individuals
Brief Title: Upper Limb Exercise Capacity: Lung Transplant vs. Healthy Controls
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: TABED 2-25-1288
Record Dates: First submitted 2025-06-25; First posted 2025-07-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: Transplant Recipient
Keywords: Lung Transplant; Upper Extremity; Exercise Capacity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Individuals
- Lung Transplant Recipients

SUMMARY:
Lung transplantation is a surgical intervention for end-stage lung diseases (e.g., COPD, cystic fibrosis, idiopathic pulmonary fibrosis). While post-transplant pulmonary function improves, peak exercise capacity remains 40-60% lower than age-matched healthy individuals due to factors like muscle weakness, reduced aerobic capacity, and immunosuppressive therapy. Although lower extremity rehabilitation is common, upper extremity (UE) function is often overlooked despite its impact on quality of life (QoL) and activities of daily living (ADLs). The 6-Minute Pegboard and Ring Test (6PBRT) evaluates UE functional capacity but has not been studied in long-term lung transplant recipients (LTRs).

Objectives:

Primary: Compare UE exercise capacity between LTRs and healthy controls using 6PBRT.

Secondary: Investigate correlations between 6PBRT performance and pulmonary function, fatigue perception, ADLs, and QoL in LTRs.

Hypotheses:

H0: No significant difference in UE exercise capacity between LTRs and healthy individuals.

H1: Significant difference exists.

Methods:

Design: Cross-sectional study. Sample size calculated based on prior 6PBRT data (effect size: 1.10, power: 80%, α: 0.05).

Assessments:

Demographics: Age, sex, BMI, Charlson Comorbidity Index (CCI). 6PBRT: Measures UE endurance (total rings moved in 6 minutes). Vital signs (SpO₂, heart rate, Borg scale for fatigue) recorded.

LTR-specific:

Pulmonary function: FEV₁, FVC, FEV₁/FVC. Fatigue: Fatigue Severity Scale (FSS; scores ≥4 indicate severe fatigue). QoL: St. George's Respiratory Questionnaire (SGRQ; 0=best, 100=worst). ADLs: London Chest ADL Questionnaire (0-5 scale).

Expected Outcomes:

LTRs will show significantly lower 6PBRT scores vs. controls. 6PBRT performance will correlate with pulmonary function, fatigue, and QoL in LTRs.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Lung Transplant Recipients:

* Patients aged 18-70 years
* At least 3 months post-lung transplantation with no major complications
* Clinically stable with any comorbidities under control
* Willing to participate in the study
* No neurological or orthopedic conditions that may interfere with functional testing
* Sufficient cognitive level to understand and perform required tests and questionnaires

Inclusion Criteria for Healthy Controls:

* Aged 18-70 years
* Sufficient cognitive ability to understand and complete the tests
* Willing to participate in the study

Exclusion Criteria:

Exclusion Criteria for Lung Transplant Recipients:

* Single-lung transplant recipients
* Patients with orthopedic limitations
* Patients unable to cooperate or comply with study procedures
* Patients with mental disorders

Exclusion Criteria for Healthy Controls:

* Presence of cardiovascular diseases, cerebrovascular disease, dementia, chronic pulmonary diseases, moderate-to-severe liver diseases, hemiplegia, moderate or severe kidney disease, or solid tumors
* Orthopedic conditions that would prevent exercise testing Inability to cooperate or comply with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lung transplant patients who are being followed up at Bilkent City Hospital Chest Surgery Clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Upper extremity functional exercise capacity | Baseline only (single assessment, no follow-up)
  Upper Extremity Functional Capacity assessed by 6-minute pegboard and ring test (6PBRT). The 6-Minute Pegboard and Ring Test (6PBRT) assesses upper limb endurance and functional capacity. The participant moves rings between pegs on a board using alternating hands for six minutes. The total number of rings moved is recorded as the outcome

SECONDARY OUTCOMES:
Respiratory Function | Baseline only (no follow-up)
  Respiratory functions will be evaluated with Pulmonary function tests (PFTs). Pulmonary function tests (PFTs) assess lung function. Key parameters include FEV₁, FVC, and the FEV₁/FVC ratio to evaluate airflow and detect obstruction or restriction. TLC measures total lung capacity. Results will be reported in liters (L) and as a percentage of predicted normal values (based on age, sex, and height).

CONTACTS AND LOCATIONS:
Locations (1):
- Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to protect participant confidentiality and comply with local data protection regulations.

REFERENCES:
- [Result] Fuller LM, El-Ansary D, Button BM, Corbett M, Snell G, Marasco S, Holland AE. Effect of Upper Limb Rehabilitation Compared to No Upper Limb Rehabilitation in Lung Transplant Recipients: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Jul;99(7):1257-1264.e2. doi: 10.1016/j.apmr.2017.09.115. Epub 2017 Oct 16. PMID 29042172
- [Result] Cakmak A, Kocaaga E, Sonbahar-Ulu H, Inal-Ince D, Vardar-Yagli N, Calik-Kutukcu E, Saglam M, Coplu L. Upper Extremity Exercise Capacity and Activities of Daily Living in Individuals With Bronchiectasis Versus Healthy Controls. Phys Ther. 2023 Apr 4;103(4):pzad012. doi: 10.1093/ptj/pzad012. PMID 37086209